CLINICAL TRIAL: NCT04829292
Title: A Framework for Research in Emerging Adults: Stepped Care for Youth at Risk of Psychosis
Brief Title: Stepped Care for Youth at Risk of Psychosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Jean Addington, PhD, Professor, University of Calgary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ACH Foundation
Record Dates: First submitted 2021-03-29; First posted 2021-04-02 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Clinical High Risk for Developing Psychosis
MeSH Terms: interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Open treatment (Experimental): Supportive therapy followed by CBT
  Interventions: Behavioral: Supportive therapy and CBT

INTERVENTIONS:
Behavioral: Supportive therapy and CBT — In this open trial participants are first offered supportive therapy followed by CBT

SUMMARY:
The study will recruit 60 young people who meet established criteria for being at clinical high risk for psychosis. They will be offered a range of psychological interventions starting with the most benign treatments in different steps. At step 1 they will be offered individual or group support and if there is no improvement they will be offered more intensive CBT individual therapy or CBSST group therapy. Assessments will occur at baseline, 6,12 and 18 months

DETAILED DESCRIPTION:
In treating youth at clinical high risk of developing psychosis we have not been able to address what treatment to offer first and when to offer more intense and, ultimately, more costly treatments. The goals of achieving Precision Health objectives require that these questions be addressed through research.

The overall aim is to determine the most effective and efficient way to offer active and maintenance treatment resources for CHR youth. The first step would be to offer a range of treatments starting with the most benign as advocated in the McGorry and Hickie stage model. We will use this project to test whether clinical staging will improve prediction of prognosis and result in improved matching of treatment. The specific objectives of this project are: (1) to determine which and what proportion of participants would remit (i) within the first 1-2 months of treatment, (ii) after a brief supportive therapy, (iii) after longer term, focused psychological interventions such as CBT, CBSST and family intervention and (iv) how many make use of medications; (2) to determine adherence of CHR individuals to different treatments; and (3) to determine the need for maintenance treatment. To assess these objectives the following outcomes will be determined:

1. Improvement of Attenuated Psychotic Symptoms
2. Improved social functioning as rated by Global: Social Functioning
3. Percentage of the sample that demonstrate either symptomatic or functional improvement after Step 1 treatments and do not require to move to Step 2 treatments.
4. Percentage of sample that move to Step 2 Treatments and the percentage that achieve improvement in either symptoms or functioning.
5. Percentage of participants allocated to a given treatment that adhere to the treatment.

Participants will be between ages 12 and 30. We will recruit 60 participants who meet well-established criteria for clinical high risk for psychosis based on the Structured Interview for Psychosis-Risk Syndromes (SIPS).

Assessments will be conducted at baseline and 2, 6, 12, and 18 months after baseline. Assessments consist of clinical assessments. Clinical raters will be experienced raters and will be trained on all clinical measures and routine reliability checks will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Meeting SIPS criteria for clinical high risk for psychosis

Exclusion Criteria:

* meeting criteria for any current or past axis I psychotic disorder, IQ less than 70, or past or current history of a clinically significant central nervous system disorder.

Ages: 12 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Scale of Psychosis Risk Symptoms | Baseline and 18 months
  Individuals' clinical symptoms will be measured using scores on positive symptoms on the SOPS.

SECONDARY OUTCOMES:
Global Functioning Scale: Social and Role | Baseline and 18 months
  Clinical rating scales to assess if there are changes in social and role functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Jean M Addington, PhD, Principal Investigator — University of Calgary
Locations (1):
- Mathison Centre for Research and Education, University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No